CLINICAL TRIAL: NCT00263276
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 2 Trial to Evaluate the Safety and Efficacy of BMS-512148 as Monotherapy in Subjects With Type 2 Diabetes Mellitus Who Are Treatment Naive And Have Inadequate Glycemic Control on Diet and Exercise
Brief Title: A Trial of BMS-512148 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-008
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Arm 1 (Experimental)
  Interventions: Drug: dapagliflozin
- Arm 2 (Experimental)
  Interventions: Drug: dapagliflozin
- Arm 3 (Experimental)
  Interventions: Drug: dapagliflozin
- Arm 4 (Experimental)
  Interventions: Drug: dapagliflozin
- Arm 5 (Experimental)
  Interventions: Drug: dapagliflozin
- Arm 6 (Placebo Comparator)
  Interventions: Drug: placebo
- Arm 7 (Active Comparator)
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: dapagliflozin — Tablets, Oral, 2.5 mg, Once daily, 12 weeks.
  Arms: Arm 1
Drug: dapagliflozin — Tablets, Oral, 5 mg, Once daily, 12 weeks.
  Arms: Arm 2
Drug: dapagliflozin — Tablets, Oral, 10 mg, Once daily, 12 weeks.
  Arms: Arm 3
Drug: dapagliflozin — Tablets, Oral, 20 mg, Once daily, 12 weeks.
  Arms: Arm 4
Drug: dapagliflozin — Tablets, Oral, 50 mg, Once daily, 12 weeks.
  Arms: Arm 5
Drug: placebo — Tablets, Oral, 0 mg, Once daily, 12 weeks.
  Arms: Arm 6
Drug: metformin — Tablets, Oral, >/= 1500 mg, Once daily, 12 weeks.
  Arms: Arm 7

SUMMARY:
The purpose of this clinical research study is to learn if BMS-512148 is effective in controlling blood sugar levels as determined by HbA1c and fasting plasma glucose in patients who have been diagnosed with Type 2 diabetes. Patients should first try to control their diabetes with diet and exercise and should not have previously been treated for their diabetes (very short periods of time are acceptable). The safety of BMS512148 will also be studied

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes mellitus with inadequate glycemic control on diet and exercise. HbA1c >= 7% and <=10%.
* Patient either has not been previously treated with antihyperglycemic medication or has been treated for <30 days since diagnosis and has received less than 3 consecutive doses or 7 non-consecutive doses in the last 30 days.
* C-peptide > 1.0 ng/ml
* Body Mass Index <= 40 kg/m2
* Serum creatinine < 1.5 mg/dL for men or < 1.4 mg/dL for women.
* No overt proteinuria (microalbumin/creatinine ratio must be <300 mg/g

Exclusion Criteria:

* Unstable renal disease
* Patients with significant liver disease including chronic active hepatitis
* Within the last 6 months has had any of the following cardiovascular event: myocardial infarction, unstable angina, unstable CHF,NYHA Class III or IV CHF, TIA, unstable arrhythmia or cardiac revascularization surgery.
* Subjects with clinically significant anemia

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in HbA1c compared to placebo. | at 12 weeks

SECONDARY OUTCOMES:
Mean change from baseline in fasting plasma glucose, evaluate proportion of subjects who achieve a therapeutic response (HbA1c <7%); change from baseline in urinary glucose excretion | at Weeks 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (144):
- United States (111):
  - Local Institution, Bayou La Batre, Alabama
  - Local Institution, Birmingham, Alabama
  - Local Institution, Huntsville, Alabama
  - Local Institution, Mobile, Alabama
  - Local Institution, Chandler, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Fayetteville, Arkansas
  - Local Institution, Hot Springs, Arkansas
  - Local Institution, Beverly Hills, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Gatos, California
  - Local Institution, Mission Viejo, California
  - Local Institution, Orange, California
  - Local Institution, Redondo Beach, California
  - Local Institution, San Diego, California
  - Local Institution, Torrance, California
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Boynton Beach, Florida
  - Local Institution, Brandon, Florida
  - Local Institution, Delray Beach, Florida
  - Local Institution, Holly Hill, Florida
  - Local Institution, Jacksonville, Florida
  - Local Instiuttion, Jacksonville, Florida
  - Local Institution, New Port Richey, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, Ormond Beach, Florida
  - Local Institution, Augusta, Georgia
  - Local Institution, Blue Ridge, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Lafayette, Indiana
  - Local Institution, Arkansas City, Kansas
  - Local Institution, Baton Rouge, Louisiana
  - Local Institution, Columbia, Maryland
  - Local Institution, Elkton, Maryland
  - Local Institution, Sudbury, Massachusetts
  - Local Institution, Worcester, Massachusetts
  - Local Institution, Dearborn, Michigan
  - Local Institution, Royal Oak, Michigan
  - Local Institution, Brooklyn Center, Minnesota
  - Local Insitution, Edina, Minnesota
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Hattiesburg, Mississippi
  - Local Institution, Jackson, Mississippi
  - Local Institution, Chesterfield, Missouri
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Scottsbluff, Nebraska
  - Local Institution, North Las Vegas, Nevada
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Los Alamos, New Mexico
  - Local Institution, Albany, New York
  - Local Institution, Bronxville, New York
  - Local Institution, Camillus, New York
  - Local Institution, Cooperstown, New York
  - Local Instiution, New Hyde Park, New York
  - Local Institution, West Seneca, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, High Point, North Carolina
  - Local Institution, Morehead City, North Carolina
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Akron, Ohio
  - Local Institution, Beachwood, Ohio
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Dayton, Ohio
  - Local Institution, Mogadore, Ohio
  - Local Institution, Newark, Ohio
  - Local Institution, Zanesville, Ohio
  - Local Institution, Bethany, Oklahoma
  - Local Institution, Yukon, Oklahoma
  - Local Institution, Bend, Oregon
  - Local Institution, Eugene, Oregon
  - Local Institution, Hillsboro, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Bensalem, Pennsylvania
  - Local Institution, Feasterville, Pennsylvania
  - Local Institution, Levittown, Pennsylvania
  - Local Institution, Morrisville, Pennsylvania
  - Local Institution, Reading, Pennsylvania
  - Local Institution, Cumberland, Rhode Island
  - Local Institution, Johnston, Rhode Island
  - Local Institution, Anderson, South Carolina
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Summerville, South Carolina
  - Local Institution, Taylors, South Carolina
  - Local Institution, Rapid City, South Dakota
  - Local Institution, Memphis, Tennessee
  - Local Institution, Nashville, Tennessee
  - Local Institution, Selmer, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Bellaire, Texas
  - Local Institution, Bryan, Texas
  - Local Institution, El Paso, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Irving, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Burke, Virginia
  - Local Institution, Hampton, Virginia
  - Local Institution, Norfolk, Virginia
  - Local Institution, Richmond, Virginia
  - Local Institution, Virginia Beach, Virginia
  - Local Institution, Edmonds, Washington
  - Local Institution, Renton, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Vancouver, Washington
  - Local Institution, Milwaukee, Wisconsin
  - Local Institution, West Allis, Wisconsin
- Canada (24):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Langley, British Columbia
  - Local Institution, Surrey, British Columbia
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local institution, Bathurst, New Brunswick
  - Local Institution, Moncton, New Brunswick
  - Local Institution, Saint John's, New Brunswick
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Corunna, Ontario
  - Local Institution, Etobicoke, Ontario
  - Local Institution, Kitchener, Ontario
  - Local Institution, Newmarket, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Drummondville, Quebec
  - Local Institution, Granby, Quebec
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Rimouski, Quebec
  - Local Institution, Saint-Léonard, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Mexico (6):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Durango, Durango
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
- Puerto Rico (3):
  - Local Institution, Caguas
  - Local Institution, Manatí
  - Local Institution, San Juan

REFERENCES:
- [Derived] Mellander A, Billger M, Johnsson E, Traff AK, Yoshida S, Johnsson K. Hypersensitivity Events, Including Potentially Hypersensitivity-Related Skin Events, with Dapagliflozin in Patients with Type 2 Diabetes Mellitus: A Pooled Analysis. Clin Drug Investig. 2016 Nov;36(11):925-933. doi: 10.1007/s40261-016-0438-3. PMID 27461213
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924
- [Derived] List JF, Woo V, Morales E, Tang W, Fiedorek FT. Sodium-glucose cotransport inhibition with dapagliflozin in type 2 diabetes. Diabetes Care. 2009 Apr;32(4):650-7. doi: 10.2337/dc08-1863. Epub 2008 Dec 29. PMID 19114612
- See also: MB102-008 _CSR_synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3632&filename=MB102-008%20_CSR_synopsis.pdf